CLINICAL TRIAL: NCT06601660
Title: Effect of Combined Physical Training At Different Times of the Day on Muscle and Adipose Tissue Remodeling, Metabolism and Physical Performance in Female Mice and Women with Obesity
Brief Title: Metabolic Investigation, Physical Performance, Physical Training At Different Times of the Day in Obese Women
Acronym: MOT-time
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of Minas Gerais (Other)
Collaborators: Federal University of Minas Gerais (Other); University of Sao Paulo (Other); Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Camila Fernanda Costa e Cunha Moraes Brandao, Professor, State University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE-59429722.1.0000.5115; APQ-02960-22 (Other Grant/Funding Number: FAPEMIG-Minas Gerais State Research Support Foundation)
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-09

CONDITIONS: Obesity Type I and II; Obesity and Overweight
Keywords: Circadian rhythm; Adipocytes; Insulin resistance; Carbohydrate metabolism; Lipid metabolism
MeSH Terms: conditions — Obesity; Overweight; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Using the randomization function of Microsoft Excel software, participants (n = 60) will be allocated into 3 experimental groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Experimental): Women who will be assessed in the morning period from 7 am to 10 am and in the evening from 6 pm to 9 pm, who will not receive intervention with combined physical training.
  Interventions: Other: No intervention
- Morning Physical Training (Experimental): Women who will perform the combined physical training at morning from 7 am to 10 am.
  Interventions: Behavioral: Morning Physical Training
- Night Physical Training (Experimental): Women who will perform the combined physical training at night from 6 pm to 9 pm.
  Interventions: Behavioral: Night Physical Training

INTERVENTIONS:
Behavioral: Morning Physical Training — A group of women who will perform the combined physical training (CPT) at morning from 7 am to 10 am, for 8 weeks and a frequency of 3 times per week (total = 24 sessions) with strength exercises and aerobic endurance exercises, performed in combination. In weeks 1 and 2, the strength training protocol will be performed with 2 sets of 16-20 maximum repetitions (RM). During weeks 3 to 5 with 12-16 RM. In weeks 6 to 8, 4 sets of 8-12 RM, with rests of 60s (weeks 1 and 2), 90s (weeks 3 to 5) and 105s (weeks 6 to 8). The minimum frequency is 90% of the training sessions. With the aerobic resistance protocol, there will be a gradual progression of the duration (volume) of the exercise (from 20 to 30 minutes per training session) and intensity (from 65% to 75% of HRres). In the first two weeks of training, participants will train at an intensity of 65% of HRres during weeks 3 to 5, at 70% of HRres in weeks 6 to 8, the intensity will reach 75% of HRres.
  Arms: Morning Physical Training
Behavioral: Night Physical Training — A group of women who will perform the combined physical training (CPT) at morning from 6 pm to 9 pm, for 8 weeks and a frequency of 3 times per week (total = 24 sessions) with strength exercises and aerobic endurance exercises, performed in combination. In weeks 1 and 2, the strength training protocol will be performed with 2 sets of 16-20 maximum repetitions (RM). During weeks 3 to 5 with 12-16 RM. In weeks 6 to 8, 4 sets of 8-12 RM, with rests of 60s (weeks 1 and 2), 90s (weeks 3 to 5) and 105s (weeks 6 to 8). The minimum frequency is 90% of the training sessions. With the aerobic resistance protocol, there will be a gradual progression of the duration (volume) of the exercise (from 20 to 30 minutes per training session) and intensity (from 65% to 75% of HRres). In the first two weeks of training, participants will train at an intensity of 65% of HRres during weeks 3 to 5, at 70% of HRres in weeks 6 to 8, the intensity will reach 75% of HRres.
  Arms: Night Physical Training
Other: No intervention — Group of women who will not receive intervention with combined physical training, but will be evaluated before and after 8 weeks, and monitored, without any intervention with physical exercise.
  Arms: Control

SUMMARY:
Obesity is a disease characterized by the accumulation of adipose tissue, which is multifactorial and can be caused by environmental, social, behavioral, biological and genetic issues, and affects people health and well-being. In this sense, it is still difficult to maintain an effective treatment for obesity, since currently in Brazil, 24% of the population is obese and 61% is overweight. Physical exercise is considered a component that promotes numerous benefits to the human body, by releasing molecules through muscle contraction that will travel throughout the body as a whole, resulting in benefits such as increased energy expenditure and, consequently, improved physical performance, which will influence a person&amp;amp;#39;s daily activities. However, the effects of physical exercise depend on some factors, such as the time and duration of the practice. In addition, the changes that occur in the body can be influenced by the time of day. Likewise, it is known how important it is to maintain adequate sleep duration at night. It is possible that the time of day when exercise is practiced influences the responses that occur in the human body. To understand this fact, obese women will undergo combined physical training (strength and aerobic exercises) performed in the morning and evening. The aim is to better understand the time of day for controlling the metabolism of obese people. And, if there is a time when people perform better in daily activities.

Therefore, the objective of this clinical trial is to evaluate whether the time of day influences the responses to combined physical training in the modulation of energy metabolism and its biochemical markers in obese women. The main questions to be answered are:

1. Can combined physical training (CPT) performed at night have different metabolic responses than CPT in the morning?
2. Can cardiopulmonary and muscular strength performance have different magnitudes of responses to CPT performed at different times of the day?
3. Can combined physical training (CPT) in the evening (NOT) compared to the morning (MAT) period cause more marked physiological adaptations, improving metabolic control in women with obesity?

DETAILED DESCRIPTION:
Obesity is a chronic, non-communicable, neuroendocrine and nutrimetabolic disease with multifactorial development, which results in a positive energy balance and excessive accumulation of adipose tissue. Characteristics of its metabolic profile include changes in mitochondrial architecture and in the secretion of hormones, such as insulin, which controls glucose metabolism. In obese individuals, adipocytes can undergo hypertrophy and hyperplasia processes, inducing low-grade inflammation. Conventional treatment for obesity consists of a hypocaloric diet combined with increased physical activity aimed at achieving a negative energy balance. However, the failure of these measures has highlighted the need for metabolic studies and studies of factors that may influence non-pharmacological treatments, such as physical training.

Physical training can improve the lipid profile of obesity, reducing cholesterol, trimethylamine N-oxide and sphingolipids, which are associated with risk factors for cardiovascular morbidity caused by obesity. An intervention with combined physical training (CPT) for 8 weeks can reduce waist circumference and increase maximum oxygen consumption in women with obesity. This approach can improve physiological functions that are altered due to obesity, such as hormonal control and bioenergetic efficiency, impacting physical fitness, regardless of weight loss. These improvements may arise depending on the configuration of the training load components, such as frequency, intensity, volume, repetition duration, pause and total session time, since it is a modifiable aspect and its manipulation provides different physiological responses.

In this sense, another factor to be considered is the circadian rhythm, which acts on metabolic regulation, and considering its functions it is assumed that it can influence the treatment of metabolic disorders, such as obesity, and physical performance. It is a biological event in which organisms go through the sleep-wake cycle, characterized by a 24-hour period that includes variations in physiological functions such as body temperature, sleep, physical activity, mood and cognition.

There are different sleep patterns and times for performing daily activities. Chronotype is a terminology that refers to the individual expression of circadian rhythmicity, a factor that is related to preferences for sleep time and duration, diet, and physical activity patterns, including exercise. Chronotype can be classified as: morning, intermediate, and evening. Based on this information, the circadian rhythm has been suggested as an influencer on responses to physical training. This biological clock can be impaired in people with metabolic disorders, such as obesity, while physical training can help regulate this clock. Several studies in humans and rodents have revealed that variables such as skeletal muscle strength and capacity demonstrate significant differences throughout the day. Therefore, this study hypothesizes that combined physical training, in the evening (NOT), compared to the morning (MAT), will cause more marked physiological adaptations, improving metabolic control, in female mice and women with obesity.

Thus, the general objective of the study will be to evaluate the effects of Combined Physical Training (CPT) performed in the morning versus evening on the remodeling of muscle and adipose tissue, metabolism and physical performance in women with obesity.

While the specific objectives:

1. To evaluate in women with obesity, before, during and after the intervention with morning TFC and evening TFC: 1.1. Body composition and body thermography; 1.2. Resting energy expenditure and oxidation of substrates (carbohydrates and lipids); 1.3. Food consumption; 1.4. Physical performance (muscular and aerobic strength); 1.5. Behavioral measures of sleep (sleep duration; sleep latency; habitual sleep duration and efficiency; circadian sleep quality and typology; daytime sleepiness); 1.6. Plasma metabolome by UPLC-MS. 1.7. Hormone levels in peripheral blood (cortisol, melatonin, corticotropin-releasing hormone - CRH, and adrenocorticotropic hormone - ACTH); 1.8. The level and phase of gene expression of the circadian cycle in peripheral blood (BMAL1, CLOCK, Cry1 and 2, Per1-3) and of energy metabolism in peripheral blood (PGC-1α, PPARγ, PPARα, NR1D1); 1.9. Verify the concentration of anti- and pro-inflammatory cytokines and myokines in peripheral blood (IL-1, IL-6, TNF-α, IL-10, IL-15 irisin, adiponectin, BNDF);

Therefore, this is an exploratory, prospective and longitudinal study, which will be carried out at the Laboratory of Research in Metabolism, Physiology and Physical Exercise of the State University of Minas Gerais, Divinópolis unit, Minas Gerais, Brazil. The sample size calculation was performed based on an equation. To perform the calculation, the chosen variable was physical performance, and data from the work of Bruggisser, was used as a source. The significance level adopted was 5%, the test power was 90%, the standard deviation was 0.80 W/kg and the difference to be detected was 0.51 W/kg. The calculation showed the need for 10 participants in each experimental group, assuming a possible loss of 20% throughout the study, the sample will consist of 12 participants per group, totaling 36 individuals of the biological female sex.

The study will last a total of 12 weeks. After verifying whether the people who have shown interest meet the inclusion criteria, they will undergo a period of anthropometric assessments, body composition, energy metabolism, blood sample collection, familiarization with the training protocol and physical tests, 2 weeks before the TFC intervention. After the TFC intervention, which will last 8 weeks and be performed 3 times a week, the same series of assessments and physical tests will be repeated for 2 weeks. Also, throughout the study, food consumption will be monitored through 24-hour recalls, and participants will be advised not to change their usual diet.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 20 and 45 years
* not practicing physical exercise
* body mass index between 30 and 39.9 kg/m²
* without any positive response when filling out the risk stratification questionnaire

Exclusion Criteria:

* Cardiovascular comorbidity
* joint and neuromuscular injuries
* diseases that affect visual and auditory functions
* disorders related to the sleep and wake cycle
* dependent on the use of psychoactive drugs
* drug treatment that influences sleep
* drug weight loss treatments
* previous bariatric surgery
* illness during the project period
* night shift workers
* attendance of 90% of the intervention with physical training

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Metabolomics | 7 months
  Blood samples will be collected before and after the eight weeks of intervention with combined physical training for analysis of the plasma metabolome, using the UPLC-MS metabolomics method.
Plasma glucose | 4 months
  Blood samples will be collected before and after the eight weeks of intervention with combined physical training for analysis of the concentration of the plasma Glucose.
Lipid profile | 4 months
  Blood samples will be collected before and after the eight weeks of intervention with combined physical training for analysis of the concentration of the Lipid profile: total cholesterol, triglycerides and lipoproteins.
Hormones | 4 months
  Blood samples will be collected before and after the eight weeks of intervention with combined physical training for analysis of the concentration of the hormones: cortisol, melatonin, corticotropin-releasing hormone (CRH) and adrenocorticotropic hormone (ACTH), insulin, growth hormone;
Genes expression | 4 months
  Blood samples will be collected before and after the eight weeks of intervention with combined physical training for analysis of the concentration of the gene expression:
  * Level and phase of gene expression and circadian rhythm protein: BMAL1, Per1 and RevErba;
  * Gene expression of energy metabolism: PGC-1a, PPARa, NR1D1
Cytokines | 4 months
  Blood samples will be collected before and after the eight weeks of intervention with combined physical training for analysis of the concentration of the Anti-inflammatory cytokines and myokines: IL-1, IL-6, IL-15, irisin, BNDF;

SECONDARY OUTCOMES:
Thermographic response | 3 months
  Tissue temperature will be assessed by a themographic camera, before and after the eight weeks of intervention with combined physical training, with the following interest regions: supraclavicular, subscapular, abdomen, forehead, hand and back.
Indirect calorimetry | 3 months
  Indirect Calorimetry: The use of gas analyzers will allow the measurement of oxygen consumption, and carbon dioxid production to calculate the resting metabolic rate, carbohydrate and lipids oxidation, and peak oxygen consumption.
  They will be evaluated before and after the intervention with combined physical training.
anthropometric measurements | 3 months
  body weight (kg) and body height (cm) will be assessed to determine the body mass index, before and after the intervention.
Multifrequency bioimpedance | 3 months
  will be assessed using multifrequency tetrapolar bioelectrical impedance (BIA) (1-1000 kHz) to measure body composition (body fat, fat-free mass, muscle mass, body water), before and after the intervention.
Dual x-ray absorptiometry | 3 months
  The mineral bone content, composition of free fat mass, lean mass, muscle mass, fat mass will all be assessed by dual x-ray absorptiometry, before and after the intervention.
cardiopulmonary fitness | 3 months
  The cardiopulmonary fitness will be evaluated in two days, being one at morning (7-10 am) and another at night (6-9 pm), before and after the intervention.
  An ergometric test with indirect calorimetry will be performed to analyze maximum oxygen consumption.
Strength performance | 3 months
  The strength performance will be evaluated in two days by 1RM test, being one at morning (7-10 am) and another at night (6-9 pm), before and after the intervention.
Blood pressure monitoring | 3 month
  The blood pressure ( systolic and diastolic) will be evaluated during intervention, by sphygmomanometer and stethoscope.
Sleep Quality Index | 3 months
  Participants will be assessed using the following questionnaires Pittsburgh Sleep Quality Index, before and after intervention.
  The instrument is divided into seven components on sleep subjectivity of the current month
Excessive daytime sleepiness | 3 months
  Participants will be assessed, before and after intervention, using the following questionnaire Epwort Sleepiness, instrument to assess excessive daytime sleepiness (EDS). Measurements above 10 on the Epworth scale are associated with sleep disturbances.
Morningness-Eveningness questionnaire | 3 months
  Participants will be assessed using the following questionnaire, before and after intervention, by Morningness-Eveningness, to determine participants' preferences.
Behavioral of sleep | 3 months
  Participants will be assessed using an actigraph (Condor Instruments) will be used, which is a wristwatch specifically designed to accurately measure activity, light and temperature on the wrist and is the ideal tool for researchers and physicians in the fields of chronobiology and sleep medicine.
Food intake | 3 months
  The food intake standart of each subject will be analyzed by a nutritionist using a 24 hours food recall (24fr) Five Step Multiple Pass method. The full amount of 24fr will be thirteen (13) for each participant, being three (3) on the first week of the study, two (2) on the physical test week pre-intervention, three (3) during the intervention, two (2) on the physical test week post-intervention, and three (3) on the last week of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Research Metabolism, Physiology and Exercise, Divinópolis, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sasaki H, Hattori Y, Ikeda Y, Kamagata M, Iwami S, Yasuda S, Tahara Y, Shibata S. Forced rather than voluntary exercise entrains peripheral clocks via a corticosterone/noradrenaline increase in PER2::LUC mice. Sci Rep. 2016 Jun 8;6:27607. doi: 10.1038/srep27607. PMID 27271267
- [Background] Kim HK, Radak Z, Takahashi M, Inami T, Shibata S. Chrono-exercise: Time-of-day-dependent physiological responses to exercise. Sports Med Health Sci. 2022 Nov 30;5(1):50-58. doi: 10.1016/j.smhs.2022.11.003. eCollection 2023 Mar. PMID 36994180
- [Background] Horne JA, Ostberg O. Individual differences in human circadian rhythms. Biol Psychol. 1977 Sep;5(3):179-90. doi: 10.1016/0301-0511(77)90001-1. PMID 922076
- [Background] Takahashi M, Tahara Y, Tsubosaka M, Fukazawa M, Ozaki M, Iwakami T, Nakaoka T, Shibata S. Chronotype and social jetlag influence human circadian clock gene expression. Sci Rep. 2018 Jul 5;8(1):10152. doi: 10.1038/s41598-018-28616-2. PMID 29976939
- [Background] Bass J, Takahashi JS. Circadian integration of metabolism and energetics. Science. 2010 Dec 3;330(6009):1349-54. doi: 10.1126/science.1195027. PMID 21127246
- [Background] Chaix A, Panda S. Timing tweaks exercise. Nat Rev Endocrinol. 2019 Aug;15(8):440-441. doi: 10.1038/s41574-019-0229-z. PMID 31217576
- [Background] Gabriel BM, Zierath JR. Circadian rhythms and exercise - re-setting the clock in metabolic disease. Nat Rev Endocrinol. 2019 Apr;15(4):197-206. doi: 10.1038/s41574-018-0150-x. PMID 30655625
- [Background] Boukelia B, Gomes EC, Florida-James GD. Diurnal Variation in Physiological and Immune Responses to Endurance Sport in Highly Trained Runners in a Hot and Humid Environment. Oxid Med Cell Longev. 2018 May 9;2018:3402143. doi: 10.1155/2018/3402143. eCollection 2018. PMID 29861827
- [Background] Mirzaei K, Xu M, Qi Q, de Jonge L, Bray GA, Sacks F, Qi L. Variants in glucose- and circadian rhythm-related genes affect the response of energy expenditure to weight-loss diets: the POUNDS LOST Trial. Am J Clin Nutr. 2014 Feb;99(2):392-9. doi: 10.3945/ajcn.113.072066. Epub 2013 Dec 11. PMID 24335056
- [Background] Conceitos da calorimetria indireta sobre distúrbios metabólicos: uma revisão narrativa. Concepts of indirect calorimetry on metabolic dis
- [Background] Bondia-Pons I, Maukonen J, Mattila I, Rissanen A, Saarela M, Kaprio J, Hakkarainen A, Lundbom J, Lundbom N, Hyotylainen T, Pietilainen KH, Oresic M. Metabolome and fecal microbiota in monozygotic twin pairs discordant for weight: a Big Mac challenge. FASEB J. 2014 Sep;28(9):4169-79. doi: 10.1096/fj.14-250167. Epub 2014 May 20. PMID 24846387
- [Background] Lee JH, Park A, Oh KJ, Lee SC, Kim WK, Bae KH. The Role of Adipose Tissue Mitochondria: Regulation of Mitochondrial Function for the Treatment of Metabolic Diseases. Int J Mol Sci. 2019 Oct 4;20(19):4924. doi: 10.3390/ijms20194924. PMID 31590292
- [Background] Uranga RM, Keller JN. The Complex Interactions Between Obesity, Metabolism and the Brain. Front Neurosci. 2019 May 24;13:513. doi: 10.3389/fnins.2019.00513. eCollection 2019. PMID 31178685
- [Background] Kahn CR, Wang G, Lee KY. Altered adipose tissue and adipocyte function in the pathogenesis of metabolic syndrome. J Clin Invest. 2019 Oct 1;129(10):3990-4000. doi: 10.1172/JCI129187. PMID 31573548
- [Background] Bruggisser F, Knaier R, Roth R, Wang W, Qian J, Scheer FAJL. Best Time of Day for Strength and Endurance Training to Improve Health and Performance? A Systematic Review with Meta-analysis. Sports Med Open. 2023 May 19;9(1):34. doi: 10.1186/s40798-023-00577-5. PMID 37208462
- [Background] Tabela Brasileira de Composição de Alimentos - TACO
- [Background] Blanton CA, Moshfegh AJ, Baer DJ, Kretsch MJ. The USDA Automated Multiple-Pass Method accurately estimates group total energy and nutrient intake. J Nutr. 2006 Oct;136(10):2594-9. doi: 10.1093/jn/136.10.2594. PMID 16988132
- [Background] La Scala Teixeira CV, Caranti DA, Oyama LM, Padovani RDC, Cuesta MGS, Moraes ADS, Cerrone LA, Affonso LHL, Gil SDS, Dos Santos RVT, Gomes RJ. Effects of functional training and 2 interdisciplinary interventions on maximal oxygen uptake and weight loss of women with obesity: a randomized clinical trial. Appl Physiol Nutr Metab. 2020 Jul;45(7):777-783. doi: 10.1139/apnm-2019-0766. Epub 2020 Jan 23. PMID 31971832
- [Background] Brandao CFC, Krempf M, Giolo de Carvalho F, Aguesse A, Junqueira-Franco MVM, Batitucci G, de Freitas EC, Noronha NY, Rodrigues GDS, Junqueira GP, Borba DA, Billon-Crossouard S, Croyal M, Marchini JS. Sphingolipid and Trimethylamine-N-Oxide (TMAO) Levels in Women with Obesity after Combined Physical Training. Metabolites. 2024 Jul 23;14(8):398. doi: 10.3390/metabo14080398. PMID 39195494
- [Background] Brandao CFC, de Carvalho FG, Souza AO, Junqueira-Franco MVM, Batitucci G, Couto-Lima CA, Fett CA, Papoti M, Freitas EC, Alberici LC, Marchini JS. Physical training, UCP1 expression, mitochondrial density, and coupling in adipose tissue from women with obesity. Scand J Med Sci Sports. 2019 Nov;29(11):1699-1706. doi: 10.1111/sms.13514. Epub 2019 Jul 22. PMID 31282585
- [Background] UCP2 expression is negatively correlated with and body fat mass after combined physical training: a pilot study
- See also: American College of Sports Medicine position stand. Progression models in resistance training for healthy adults — https://doi.org/10.1249/mss.0b013e3181915670
- See also: ACSM's Guidelines for Exercise Testing and Prescription, 11th edition — https://www.acsm.org/education-resources/books/guidelines-exercise-testing-prescription
- See also: Tabela para Avaliação do Consumo Alimentar em Medidas Caseiras 4a edição — https://nutrisaude14.wordpress.com/wp-content/uploads/2014/08/tabela-de-medidas-caseiras.pdf
- See also: Ciência do treinamento desportivo — https://pt.scribd.com/document/125125672/Ciencia-do-Treinamento-Desportivo-Zakharov
- See also: MUSCULAÇÃO: Variáveis Estruturais Programas de Treinamento Força Muscular — https://www.galaxcms.com.br/up_crud_comum/4107/MusculacaoVariaveisEstruturais3edicao-20230714120253.pdf